CLINICAL TRIAL: NCT05259852
Title: Development of A Navigation Pilot Intervention to Address the Double Burden of Food Insecurity and Tobacco Use in the Clinical Setting
Brief Title: An Intervention to Promote Smoking Cessation Among Adults With Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jin Kim-Mozeleski, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kim-MozeleskiStudy20210127
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation; Food Insecurity
MeSH Terms: conditions — Smoking Cessation | interventions — Food Assistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Assistance and Cessation Resources Navigation Plus Economic Assistance (Experimental)
  Interventions: Behavioral: Food Assistance and Cessation Resources Navigation Plus Economic Assistance
- Food Assistance and Cessation Resources Navigation (Active Comparator)
  Interventions: Behavioral: Food Assistance and Cessation Resources Navigation

INTERVENTIONS:
Behavioral: Food Assistance and Cessation Resources Navigation Plus Economic Assistance — The intervention arm involves an initial telephone call with a community health worker (CHW). The content of the call focuses on providing participants with referrals for available food assistance resources in the community and referrals for tobacco cessation services. There are two additional follow-up calls approximately 4 weeks apart, for a total of 3 CHW navigator calls over the 12-week study period. In addition, the intervention arm involves providing participants with economic assistance for food in the form of a reloadable debit card ($83 every 4 weeks for 12 weeks, for a maximum amount of $250).
  Arms: Food Assistance and Cessation Resources Navigation Plus Economic Assistance
Behavioral: Food Assistance and Cessation Resources Navigation — The comparison arm involves an initial telephone call with a community health worker (CHW). The content of the call focuses on providing participants with referrals for available food assistance resources in the community and referrals for tobacco cessation services. There are two additional follow-up calls approximately 4 weeks apart, for a total of 3 CHW navigator calls over the 12-week study period.
  Arms: Food Assistance and Cessation Resources Navigation

SUMMARY:
This is a two-arm randomized controlled study with 60 participants. The study has two aims. The first aim is to determine the feasibility and acceptability of a food assistance intervention to alleviate food insecurity during a smoking cessation attempt among low-income smokers with food insecurity. Smokers with recent food insecurity are recruited for a 12-week study that involves resources navigation for food assistance and tobacco cessation, with assessments at baseline and at 12 weeks. Participants are randomized to receive economic assistance for food in addition to resources navigation in the intervention arm, or randomized to receive resources navigation only in the control arm. The second aim is to estimate the preliminary impact of the intervention on food insecurity and tobacco cessation measures at 12 weeks.

DETAILED DESCRIPTION:
Tobacco use remains a leading cause of preventable disease, disability, and early death. National-level data show that the majority of smokers are interested in quitting and attempt to quit each year, but there are socioeconomic disparities in successfully quitting. In particular, smoking cessation can be especially hard when smokers are dealing with unmet social and health needs and areas of financial stress, which are disproportionately experienced by low-income smokers. This study extends previous research showing that food insecurity is independently associated with higher odds of smoking and can act as a barrier to quitting smoking. The study's main research question is whether alleviating food insecurity specifically during a smoking cessation attempt is helpful for increasing quitting success rates. Therefore, the study is testing a 12-week intervention to assist food-insecure smokers who are ready and willing to make a quit attempt. Beyond providing the quit assistance that smokers normally receive through healthcare providers, the research seeks to address food insecurity in the short-term by providing economic assistance for food during the quit attempt that will help to meet food needs. The study will adapt a patient navigation model in which a designated study navigator can help bridge resources and referrals related to tobacco cessation and food access, and provide economic food assistance based on individualized needs. The study will recruit 60 participants for a 12-week study, and all participants will be smokers who are ready to quit and have recently experienced food insecurity. All participants will receive quit assistance and information on local food assistance resources, and a monthly check-in from the navigator. In addition, half of the participants (n=30) will be randomly assigned to the intervention arm, and will receive economic food assistance to alleviate food insecurity during the cessation attempt. The first aim is to assess feasibility and acceptability of the intervention, and the second aim is to estimate preliminary outcomes related to smoking cessation, such as the number of quit attempts lasting 24 hours or more and the longest length of abstinence from tobacco, and reduction in food insecurity during the intervention period. By conducting this study, the investigators seek to understand whether this type of intervention is feasible to conduct, and acceptable to those who participate. The study findings will serve as the basis of future research on understanding and addressing tobacco-related and food insecurity-related health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 or older
* Current tobacco smoker, defined as having smoked daily over the past 7 days
* Willing to make a serious quit attempt in the next 30 days ("Yes" to "In the next 30 days, are you willing to try quitting smoking for at least 24 hours?")
* Considered food insecure, based on past 30-day screening using the 2-item Hunger Vital Sign, or by virtue of having visited a food pantry in the past 30 days
* Primary food shopper of household, who does half or more of the household food shopping
* A reliable telephone number and a local mailing address where participant can be reached during the duration of the study

Exclusion Criteria:

* Aged 20 or younger
* Non-smoker, or did not smoke daily over the past 7 days
* Not interested in quitting at this time, assessed by unwillingness to make a serious quit attempt in the next 30 days ("No" to "In the next 30 days, are you willing to try quitting smoking for at least 24 hours?")
* Did not recently experience food insecurity, based on past 30-day screening using the 2-item Hunger Vital Sign, or has not visited a food pantry in the past 30 days
* Not the primary food shopper of the household (does less than half of the household food shopping)
* Does not have a reliable telephone number and a local mailing address where participant can be reached during the duration of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim-Mozeleski JE, Castele MC, Nambiar P, Chagin KM, Pike Moore S, Hardy P, Cook K, Sehgal AR. A Randomized Trial to Address Food Insecurity and Promote Smoking Cessation Among Low-Income Adults. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241245275. doi: 10.1177/21501319241245275. PMID 38584453

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation
Started | 28 | 27
Completed | 25 | 19
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (15.3) | 49.9 (12.6) | 50.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 12 | 12 | 24
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Education [Count of Participants; unit: Participants]
  Did not complete high school | 3 | 3 | 6
  High school graduate or GED | 9 | 10 | 19
  Some college | 15 | 9 | 24
  College degree | 0 | 3 | 3
  More than a college degree | 1 | 2 | 3
  Prefer not to answer | 0 | 0 | 0
Annual household income [Count of Participants; unit: Participants]
  Less than $10,000 | 9 | 6 | 15
  $10,000 - $19,999 | 9 | 10 | 19
  $20,000 - $39,999 | 7 | 9 | 16
  $40,000 - $59,999 | 0 | 2 | 2
  $60,000 - $79,999 | 2 | 0 | 2
  $80,000 or higher | 0 | 0 | 0
  Prefer not to answer | 1 | 0 | 1
Marital status [Count of Participants; unit: Participants]
  Single, never married | 17 | 15 | 32
  Married or partnered | 3 | 3 | 6
  Divorced or separated | 7 | 7 | 14
  Widowed | 1 | 2 | 3
  Prefer not to answer | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of 24-hour Quit Attempts
Description: In the past 3 months, how many times did you stop using tobacco for 24 hours or more because you were trying to quit smoking?
Time Frame: 3 months
Population: Complete case analysis
Measure: Mean (Standard Deviation); unit: number of 24-hour quit attempts
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation
Number analyzed (Participants) | 25 | 19
number of 24-hour quit attempts | 2.6 (1.8) | 1.8 (1.7)

2. Primary Outcome: Longest Length of Abstinence in Days
Description: In the past 3 months, what was the longest time (in days) you went without using tobacco?
Time Frame: 3 months
Population: complete case analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation
Number analyzed (Participants) | 25 | 19
days | 18.7 (21.0) | 9.3 (15.5)

3. Primary Outcome: Level of Food Security
Description: 6-item Adult/Household Food Security Survey by the US Dept of Agriculture
Time Frame: 3 months
Population: complete case analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation
Number analyzed (Participants) | 25 | 19
Participants
  High/marginal food security | 4 | 4
  Low food security | 12 | 7
  Very low food security | 9 | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period, from the beginning to end of data collection.
Arm/Group | Food Assistance and Cessation Resources Navigation Plus Economic Assistance | Food Assistance and Cessation Resources Navigation
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT05259852/Prot_SAP_000.pdf